CLINICAL TRIAL: NCT06015074
Title: Ciprofol vs Propofol for Reducing Hypoxia Incidence in Intravenous Anesthesia During Elective Endoscopic Retrograde Cholangiopancreatography-A Randomized Double Blinded Controlled Trial.
Brief Title: Ciprofol vs Propofol for Reducing Hypoxia Incidence in ERCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: C-Anesthesia
Record Dates: First submitted 2023-06-21; First posted 2023-08-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Adverse Effect; Biliary Tract Diseases
Keywords: Ciprofol; Propofol; Intravenous Anesthesia; Elective Endoscopic Retrograde Cholangiopancreatography; Hypoxia
MeSH Terms: conditions — Biliary Tract Diseases; Hypoxia | interventions — Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Active Comparator): patients in Propofol group receive sufentanil+ propofol
  Interventions: Drug: Propofol
- Ciprofol group (Experimental): patients in Ciprofol group receive sufentanil+ ciprofol
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Propofol — patients in Propofol group receive sufentanil(0.1ug/kg)+ propofol (1.5-2mg/kg) for anesthesia induction, and continuous infusion of propofol 5mg/kg/h for anesthesia maintain.
  Other Names: Fresenius Kabi，China
  Arms: Propofol group
Drug: Ciprofol — patients in Ciprofol group receive sufentanil(0.1ug/kg)+ ciprofol(0.4-0.5mg/kg) for anesthesia induction, and continuous infusion of ciprofol 0.8mg/kg/h for anesthesia maintain.
  Other Names: Haisike，China
  Arms: Ciprofol group

SUMMARY:
Intravenous anesthesia has been widely used in endoscopic retrograde cholangiopancreatography (ERCP). In the past decade, many practices have been carried out under the propofol-based monitored anesthesia care without endotracheal intubation in patients undergoing ERCP.

Ciprofol is a newly developed intravenous anesthetic with a potency 4-5 times than that of propofol. Ciprofol seems a promising anesthetic agent for intravenous anesthesia but the evidence supported its application in ERCP is still limited.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind trial comparing the incidence of hypoxia in the propofol versus ciprofol intravenous Anesthesia. A total 136 patients will be recruited and randomly assigned to either the propofol or the ciprofol group. The primary outcome is the proportion of patients experiencing hypoxia. The secondary outcomes include: the incidence of hypotension in perioperative period; the incidence of conversion from intravenous anesthesia to general anesthesia; sedation-related procedure interruption; carbon dioxide( CO2) accumulation during operation; Patients' satisfaction with anesthesia and postoperative recovery / VAS score / incidence of nausea and vomiting; the incidence of intraoperative and postoperative adverse events, such as adverse excretion, severe hypoxemia, severe circulatory dysfunction; length of stay and mortality within 30 days after operation.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing ERCP, ASA I-III
* normal renal function
* BMI ≥ 18kg/m 2 and ≤ 30kg/m 2

Exclusion Criteria:

* Previous serious cerebrovascular accidents and other neurological diseases
* mental diseases, long-term use of drugs that affect the function of the central nervous system, benzodiazepines or opioids
* history of anesthetic allergy
* preoperative hypotension or preoperative SpO2 < 90%, or chronic respiratory failure
* patients suspected of having difficult airways
* screening for drug addiction and alcohol abuse within the first 3 months (> = 6standarddrinks/day)
* patients diagnosed with severe cardiopulmonary disease, or respiratory or respiratory diseases such as sleep apnea syndrome;
* bradycardia or atrioventricular block.
* participate in other clinical trials within 4 weeks;
* cognitive or communication abnormalities determined by the researchers;
* emergent and critical conditions during the operation;
* other conditions that the researchers believe are not suitable to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
the incidence of hypoxia | from the induction of anesthesia to the patient leaving the postanesthesia care unit，about an average of 1.5 hours
  the definition of hypoxemia: any event of SpO2 (oxygen saturation measured by pulse oximetry) < 90%

SECONDARY OUTCOMES:
the incidence of hypercapnia | 5 minutes each time（base line, 10 minutes after beginning of surgery, completion of surgery, 10 minutes after awakening）
  arterial carbon dioxide partial pressure（PaCO2）>50mmHg
the incidence of hypotension | from the induction of anesthesia to the patient leaving the postanesthesia care unit，about an average of 1.5 hours
  invasive systolic pressure<90mmHg
sedation-related procedure interruption | from the induction of anesthesia to completion of ERCP, about 30 minutes
  the incidence of interruption of procedure due to intolerance or severe adverse events
conversion from intravenous anesthesia to general anesthesia | from the induction of anesthesia to completion of ERCP, about 30 minutes
  the incidence of conversion from intravenous anesthesia to general anesthesia due to intolerance or severe adverse events
patient satisfaction score | 5 minutes
  Patients' satisfaction score is measured by patient recovery satisfaction score, from -33 the worst to 33 the best.
visual analog scale (VAS) scores | 30 seconds
  perioperative pain is measured by visual analog scale (VAS) scores，from painless score 0 to the imagined most severe pain score 10
length of stay | 2-7days
  length of stay in hospital
the incidence of postoperative adverse bile excretion | 30 days after operation
  patients with symptoms or signs of postoperative adverse bile excretion
the incidence of severe postoperative hypoxia | 30 days after operation
  patients with symptoms or signs of severe postoperative hypoxia
the incidence of severe postoperative circulatory disfunction | 30 days after operation
  patients with symptoms or signs of severe postoperative circulatory disfunction
the incidence of mortality within 30 days after operation | 30 days after operation
  mortality within 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Peiying Li, Doctor, Study Director — Clinial Research Center, Renji Hospital; Yu Weifeng, Doctor, Study Chair — Department of Anesthesiology, Renji Hospital; Zheng Li, Master, Study Director — Department of Anesthesiology, Renji Hospital; Yanhua Zhao, Doctor, Principal Investigator — Department of Anesthesiology, Renji Hospital; Yifeng Qu, Master, Principal Investigator — Department of Anesthesiology, Renji Hospital; Kun Luo, Master, Principal Investigator — Department of Anesthesiology, Renji Hospital; Guangyan Wang, Principal Investigator — Operating Room，Renji Hospital; Teng Wang, Principal Investigator — Department of Anesthesiology, Renji Hospital; Huichen Zhu, Master, Principal Investigator — Department of Anesthesiology, Renji Hospital; Jing Gao, Doctor, Principal Investigator — Clinial Research Center, Renji Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler DG, Baron TH, Davila RE, Egan J, Hirota WK, Leighton JA, Qureshi W, Rajan E, Zuckerman MJ, Fanelli R, Wheeler-Harbaugh J, Faigel DO; Standards of Practice Committee of American Society for Gastrointestinal Endoscopy. ASGE guideline: the role of ERCP in diseases of the biliary tract and the pancreas. Gastrointest Endosc. 2005 Jul;62(1):1-8. doi: 10.1016/j.gie.2005.04.015. No abstract available. PMID 15990812
- [Background] Alzanbagi AB, Jilani TL, Qureshi LA, Ibrahim IM, Tashkandi AMS, Elshrief EEA, Khan MS, Abdelhalim MAH, Zahrani SA, Mohamed WMK, Nageeb AM, Abbushi B, Shariff MK. Randomized trial comparing general anesthesia with anesthesiologist-administered deep sedation for ERCP in average-risk patients. Gastrointest Endosc. 2022 Dec;96(6):983-990.e2. doi: 10.1016/j.gie.2022.06.003. Epub 2022 Jun 9. PMID 35690151
- [Background] Cote GA, Hovis RM, Ansstas MA, Waldbaum L, Azar RR, Early DS, Edmundowicz SA, Mullady DK, Jonnalagadda SS. Incidence of sedation-related complications with propofol use during advanced endoscopic procedures. Clin Gastroenterol Hepatol. 2010 Feb;8(2):137-42. doi: 10.1016/j.cgh.2009.07.008. Epub 2009 Jul 14. PMID 19607937
- [Background] Amornyotin S, Srikureja W, Chalayonnavin W, Kongphlay S. Dose requirement and complications of diluted and undiluted propofol for deep sedation in endoscopic retrograde cholangiopancreatography. Hepatobiliary Pancreat Dis Int. 2011 Jun;10(3):313-8. doi: 10.1016/s1499-3872(11)60052-0. PMID 21669577
- [Background] Qadeer MA, Vargo JJ, Dumot JA, Lopez R, Trolli PA, Stevens T, Parsi MA, Sanaka MR, Zuccaro G. Capnographic monitoring of respiratory activity improves safety of sedation for endoscopic cholangiopancreatography and ultrasonography. Gastroenterology. 2009 May;136(5):1568-76; quiz 1819-20. doi: 10.1053/j.gastro.2009.02.004. PMID 19422079
- [Background] Vargo JJ, Zuccaro G Jr, Dumot JA, Conwell DL, Morrow JB, Shay SS. Automated graphic assessment of respiratory activity is superior to pulse oximetry and visual assessment for the detection of early respiratory depression during therapeutic upper endoscopy. Gastrointest Endosc. 2002 Jun;55(7):826-31. doi: 10.1067/mge.2002.124208. PMID 12024135
- [Background] Paspatis GA, Manolaraki MM, Vardas E, Theodoropoulou A, Chlouverakis G. Deep sedation for endoscopic retrograde cholangiopancreatography: intravenous propofol alone versus intravenous propofol with oral midazolam premedication. Endoscopy. 2008 Apr;40(4):308-13. doi: 10.1055/s-2007-995346. Epub 2007 Dec 5. PMID 18058653
- [Background] Vargo JJ, Zuccaro G Jr, Dumot JA, Shermock KM, Morrow JB, Conwell DL, Trolli PA, Maurer WG. Gastroenterologist-administered propofol versus meperidine and midazolam for advanced upper endoscopy: a prospective, randomized trial. Gastroenterology. 2002 Jul;123(1):8-16. doi: 10.1053/gast.2002.34232. PMID 12105827
- [Background] Liu Y, Yu X, Zhu D, Zeng J, Lin Q, Zang B, Chen C, Liu N, Liu X, Gao W, Guan X. Safety and efficacy of ciprofol vs. propofol for sedation in intensive care unit patients with mechanical ventilation: a multi-center, open label, randomized, phase 2 trial. Chin Med J (Engl). 2022 May 5;135(9):1043-1051. doi: 10.1097/CM9.0000000000001912. PMID 34924506
- [Background] Liu Y, Chen C, Liu N, Tong L, Nie Y, Wu J, Liu X, Gao W, Tang L, Guan X. Efficacy and Safety of Ciprofol Sedation in ICU Patients with Mechanical Ventilation: A Clinical Trial Study Protocol. Adv Ther. 2021 Oct;38(10):5412-5423. doi: 10.1007/s12325-021-01877-6. Epub 2021 Aug 21. PMID 34417990